CLINICAL TRIAL: NCT07074535
Title: CT and Endoscopic Biopsy Image-Based Deep Learning for Predicting Left Recurrent Laryngeal Nerve Lymph Node Metastasis in Esophageal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CEDREL-LNM
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Squamous Cell Cancer (SCC); Recurrent Laryngeal Nerve Palsy; Deep Learning; Postoperative Complication
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Vocal Cord Paralysis; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Left RLN lymph node （+）: Postoperative pathological results confirmed the metastasis of left recurrent laryngeal nerve lymph nodes.
- Left RLN lymph node （-）: Postoperative pathological results confirmed the negative of left recurrent laryngeal nerve lymph nodes.

SUMMARY:
The goal of this observational study is to develop a predictive model for left recurrent laryngeal nerve (RLN) lymph node metastasis using deep learning algorithms. The model will be developed using clinical data from previous esophageal cancer surgeries, including preoperative CT imaging, and histopathological images from gastroscopic biopsies. The model will also be validated through prospective clinical trials to guide the intraoperative lymph node dissection, thereby reducing postoperative risks of RLN injury.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative gastroscopic biopsy confirmed esophageal squamous cell carcinoma；
* The patient underwent esophagectomy with lymph nodes dissection along the left recurrent laryngeal nerve.

Exclusion Criteria:

* The patient's medical records are incomplete；
* The patient refused to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included were all esophageal cancer patients who received surgery and standard lymph node dissection in our hospital.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
AUROC (Area Under the Receiver Operating Characteristic Curve) | From enrollment to the end of treatment at 4 weeks
  The discriminant ability of the comprehensive evaluation model at different thresholds (positive vs. negative)

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided
Datasets and codes for the study are available from the corresponding author on reasonable request.